CLINICAL TRIAL: NCT00954642
Title: A Phase Ib, Open-Label, Dose-Escalation Study of the Safety and Pharmacology of MNRP1685A, a Human IgG1 Antibody, in Combination With Bevacizumab With or Without Paclitaxel in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study of MNRP1685A in Combination With Bevacizumab With or Without Paclitaxel in Patients With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANP4667g
Record Dates: First submitted 2009-08-05; First posted 2009-08-07 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Solid Cancers
Keywords: Solid Tumor; Locally Advanced Solid Tumor; Avastin
MeSH Terms: interventions — Bevacizumab; vesencumab; Paclitaxel

ARMS (2):
- A (Experimental)
  Interventions: Drug: bevacizumab; Drug: MNRP1685A
- B (Experimental)
  Interventions: Drug: bevacizumab; Drug: MNRP1685A; Drug: paclitaxel

INTERVENTIONS:
Drug: bevacizumab — Intravenous repeating dose
Drug: MNRP1685A — Escalating intravenous dose
Drug: paclitaxel — Intravenous repeating dose
  Arms: B

SUMMARY:
This is a Phase Ib, open-label, dose-escalation study of MNRP1685A given by intravenous (IV) infusion as therapy for locally advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Adequate hematologic and end organ function
* Evaluable disease or measurable disease per Response Evaluation Criteria In Solid Tumors (RECIST)
* Agreement to use an effective form of contraception for the duration of the study

Inclusion Criteria Unique to Arm A:

* Histologically or cytologically documented, incurable, locally advanced, or metastatic solid malignancy that has progressed on, or failed to respond to, at least one prior regimen

Inclusion Criteria Unique to Arm B:

* Histologically or cytologically documented, incurable, locally advanced, or metastatic solid malignancy; a maximum of two prior chemotherapy regimens is allowed

Exclusion Criteria:

* Any anti-cancer therapy, including chemotherapy, hormonal therapy, or radiotherapy, within 3 weeks or 5 half-lives (for systemic agents), whichever is shorter, prior to initiation of study treatment with the following exceptions: hormonal therapy with gonadotropin-releasing hormone (GnRH) agonists or antagonists for prostate cancer; herbal therapy > 1 week prior to Day 1; hormone-replacement therapy or oral contraceptives; palliative radiotherapy for bone metastases > 2 weeks prior to Day 1
* Any condition requiring full-dose anticoagulants, such as warfarin, heparin, or thrombolytics, or a filter of the inferior vena cava
* Leptomeningeal disease as a manifestation of the current malignancy
* Active infection requiring IV antibiotics
* Active autoimmune disease that is not controlled by nonsteroidal anti-inflammatory drugs, inhaled corticosteroids, or the equivalent of ≤ 10 mg/day prednisone
* Bisphosphonate therapy for symptomatic hypercalcemia
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis, or cirrhosis
* Known human immunodeficiency virus (HIV) infection
* Known primary CNS malignancy, or untreated or active CNS metastases
* Pregnancy, lactation or breast feeding
* Inadequately controlled hypertension
* History of hypertensive crisis or hypertensive encephalopathy
* History of myocardial infarction or unstable angina within 6 months prior to Day 1
* New York Heart Association (NYHA) Class II or greater CHF
* History of stroke or transient ischemic attack (TIA) within 6 months prior to Day 1
* Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Day 1
* History of hemoptysis within 1 month prior to Day 1
* Evidence of bleeding diathesis or significant coagulopathy in the absence of stable therapeutic anticoagulation
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to Day 1
* History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months prior to Day 1
* Clinical signs or symptoms of gastrointestinal obstruction or requirement for parenteral hydration, parenteral nutrition, or tube feeding because of an active gastrointestinal condition
* Evidence of abdominal free air not explained by paracentesis or recent surgical procedure
* Serious, non-healing wound, active gastrointestinal ulcer, or untreated bone fracture
* Intrathoracic lung carcinoma of squamous cell histology
* Grade ≥ 2 sensory neuropathy
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
* Known hypersensitivity to recombinant human antibodies

Exclusion Criterion Unique to Arm B:

* Known significant hypersensitivity to paclitaxel or other drugs using the vehicle cremophor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-08 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Incidence and nature of dose-limiting toxicities (DLTs) | Through study completion or early study discontinuation

SECONDARY OUTCOMES:
Pharmacokinetic (PK) parameters of MNRP1685A and bevacizumab, when appropriate, as data allow (total exposure, maximum and minimum serum concentration, clearance, and volume of distribution) | Through study completion or early study discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Brachmann, M.D., Study Director — Genentech, Inc.